CLINICAL TRIAL: NCT03544294
Title: veRy Thin Stents for Patients With Left mAIn or bifurcatioN in Real Life: the RAIN a Multicenter Study
Acronym: RAIN
Status: Completed | Type: Observational
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Collaborators: University Hospital, Zürich (Other)
Responsible Party: Principal Investigator, Fabrizio D'Ascenzo, Principal Investigator, A.O.U. Città della Salute e della Scienza
Other Study IDs: RAIN
Record Dates: First submitted 2018-05-18; First posted 2018-06-01 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Stent Restenosis; Stent Thrombosis; Left Main Coronary Artery Disease; Coronary Bifurcations; Very Thin Stents
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Group: Consecutive patients treated with very thin stents on ULM and bifurcation
  Interventions: Device: Xience alpine, ultimaster, resolute onyx, synergy

INTERVENTIONS:
Device: Xience alpine, ultimaster, resolute onyx, synergy — PCI will be performed

SUMMARY:
For permanent coronary stents, reduction of thickness of struts have become one of the most important innovation, being related to easier manipulation, reduced risk of stent thrombosis and low rate of revascularization. Consequently the investigators performed a multicenter registry enrolling all consecutive patients treated with very thin stents for ULM or bifurcation.

DETAILED DESCRIPTION:
For permanent coronary stents, reduction of thickness of struts have become one of the most important innovation, being related to easier manipulation, reduced risk of stent thrombosis and low rate of revascularization. Previous studies do not have enough power to detect potential significant difference for ULM or bifurcation lesions. Consequently the investigators performed a multicenter registry enrolling all consecutive patients treated with Biomatrix Flex, Xience Alpine, Ultimaster, Resolute Onyx and Synergy. MACE (a composite end point of death, myocardial infarction, target lesion revascularization and stent thrombosis) will be the primary end point, while its single components will be the secondary ones.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing PCI on unprotected left main or coronary bifurcation

Exclusion Criteria:

* PCI performed on other coronary vessels

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients undergoing PCI
Sampling Method: Probability Sample
Enrollment: 2800 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events (MACE) | 1 year
  Major Adverse Cardiac Events (MACE) is a composite end-point which includes: death for any cause; non fatal myocardial infarction; target lesion revascularization (TLR); in-stent thrombosis.

SECONDARY OUTCOMES:
Target Lesion revascularization (TLR) | 1 year
  The investigators defined Target Lesion Revascularization as either repeat percutaneous or surgical revascularization for a lesion anywhere within the stent or the 5-mm borders proximal or distal to the stent.
Death | 1 year
  Death for any cause (both cardiologic and non-cardiologic)
non fatal myocardial infarction | 1 year
  non fatal myocardial infarction
Target Vessel Revascularization (TVR) | 1 year
  TVR is defined as any repeat PCI in the target vessel indicating the disease progression.

CONTACTS AND LOCATIONS:
Locations (1):
- Citta della Salute, Turin, Italy

REFERENCES:
- [Derived] Choi KH, Nam CW, Bruno F, Cho YK, De Luca L, Kang J, Mattesini A, Song YB, Truffa A, Kim HS, Wanha W, Chun WJ, Gili S, Helft G, Han SH, Cortese B, Lee CH, Escaned J, Yoon HJ, Chieffo A, Hahn JY, Gallone G, Choi SH, De Ferrari G, Koo BK, Quadri G, Hur SH, D'Ascenzo F, Gwon HC, de Filippo O. Differential Prognosis of True Bifurcation Lesions According to Left Main Versus Non-Left Main Location and Treatment Strategy. J Am Heart Assoc. 2025 Feb 4;14(3):e037657. doi: 10.1161/JAHA.124.037657. Epub 2025 Feb 3. PMID 39895551
- [Derived] Choi KH, Bruno F, Cho YK, De Luca L, Song YB, Kang J, Mattesini A, Gwon HC, Truffa A, Kim HS, Wanha W, Chun WJ, Gili S, Hur SH, Helft G, Han SH, Cortese B, Lee CH, Escaned J, Yoon HJ, Chieffo A, Hahn JY, Gallone G, Choi SH, De Ferrari G, Koo BK, Quadri G, D'Ascenzo F, Nam CW, de Filippo O. Comparison of Outcomes Between 1- and 2-Stent Techniques for Medina Classification 0.0.1 Coronary Bifurcation Lesions. JACC Cardiovasc Interv. 2023 Sep 11;16(17):2083-2093. doi: 10.1016/j.jcin.2023.06.013. Epub 2023 Aug 9. PMID 37565964
- [Derived] Iannaccone M, Barbero U, De Benedictis M, Imori Y, Quadri G, Trabattoni D, Ryan N, Venuti G, Montabone A, Wojakowski W, Rognoni A, Helft G, Parma R, De Luca L, Autelli M, Boccuzzi G, Mattesini A, Templin C, Cerrato E, Wanha W, Smolka G, Huczek Z, Tomassini F, Cortese B, Capodanno D, Chieffo A, Nunez-Gil I, Gili S, Bassignana A, di Mario C, Doronzo B, Omede P, D'Amico M, Tedeschi D, Varbella F, Luscher T, Sheiban I, Escaned J, Rinaldi M, D'Ascenzo F. Comparison of bioresorbable vs durable polymer drug-eluting stents in unprotected left main (from the RAIN-CARDIOGROUP VII Study). BMC Cardiovasc Disord. 2020 May 15;20(1):225. doi: 10.1186/s12872-020-01420-5. PMID 32414330
- [Derived] Gaido L, D'Ascenzo F, Imori Y, Wojakowski W, Saglietto A, Figini F, Mattesini A, Trabattoni D, Rognoni A, Tomassini F, Bernardi A, Ryan N, Muscoli S, Helft G, De Filippo O, Parma R, De Luca L, Ugo F, Cerrato E, Montefusco A, Pennacchi M, Wanha W, Smolka G, de Lio G, Bruno F, Huczek Z, Boccuzzi G, Cortese B, Capodanno D, Omede P, Mancone M, Nunez-Gil I, Romeo F, Varbella F, Rinaldi M, Escaned J, Conrotto F, Burzotta F, Chieffo A, Perl L, D'Amico M, di Mario C, Sheiban I, Gagnor A, Giammaria M, De Ferrari GM. Impact of Kissing Balloon in Patients Treated With Ultrathin Stents for Left Main Lesions and Bifurcations: An Analysis From the RAIN-CARDIOGROUP VII Study. Circ Cardiovasc Interv. 2020 Mar;13(3):e008325. doi: 10.1161/CIRCINTERVENTIONS.119.008325. Epub 2020 Feb 27. PMID 32102566